CLINICAL TRIAL: NCT01703325
Title: Comparison of Efficacy and Safety of Psoriatic Nails Treatment Between by Intralesional 0.1%Triamcinolone Injection and Topical 0.05%Clobetasol Propionate Ointment
Brief Title: Comparison of Efficacy of Intralesional Triamcinolone Injection and Clobetasol Propionate Ointment for Psoriatic Nails
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, chanisada tuchinda, Assistant Professor, Mahidol University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Si599/2010
Record Dates: First submitted 2012-06-15; First posted 2012-10-10 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Psoriatic Nails
Keywords: Psoriatic nails; Triamcinolone injection; clobetasol propionate
MeSH Terms: interventions — Triamcinolone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- triamcinolone injection (10 mg/ml) (Active Comparator): Three finger nails are chosen from the equally average Targeted NAPSI scores which are evaluated by two independent dermatologists. Block randomization are performed to arrange such fingers into group A, B or C
  Group A: Triamcinolone injection (10 mg/ml) on 4 sites for the pathology from both nail matrix (B) and nail bed (A) or 2 sites for the pathology from either nail matrix(B) or nail bed (A) as shown in picture, the EMLA was applied before injection
  Interventions: Drug: 0.1% triamcinolone , 0.05% clobetasol propionate ointment
- Topical 0.05% clobetasol ointment (Active Comparator): Three finger nails are chosen from the equally average Targeted NAPSI scores which are evaluated by two independent dermatologists. Block randomization are performed to arrange such fingers into group A, B or C Apply Topical 0.05% clobetasol propionate ointment on the nail fold twice daily for 6 months
  Interventions: Drug: 0.1% triamcinolone , 0.05% clobetasol propionate ointment
- Controlled group (No Intervention): Three finger nails are chosen from the equally average Targeted NAPSI scores which are evaluated by two independent dermatologists. Block randomization are performed to arrange such fingers into group A, B or C Controlled group

INTERVENTIONS:
Drug: 0.1% triamcinolone , 0.05% clobetasol propionate ointment — Three finger nails are chosen from the equally average NAPSI scores which are evaluated by two independent dermatologists. Block randomization are performed to arrange such fingers into group A, B or C
  * Group A: Triamcinolone injection (10 mg/ml) on 4 sites for the pathology from both nail matrix (B) and nail bed (A) or 2 sites for the pathology from either nail matrix(B) or nail bed (A) as shown in picture, the EMLA was applied before injection
  * Group B: Apply Topical 0.05% clobetasol propionate ointment (Dermovate®) on the nail fold twice daily for 6 months
  * Group C: Controlled group
  Other Names: Dermovate ointment
  Arms: Topical 0.05% clobetasol ointment; triamcinolone injection (10 mg/ml)

SUMMARY:
Psoriatic nails can significantly affect a quality of life of patients. Psoriasis affects both nail matrix and nail bed. Pitting, leukonychia and red spots in lunula indicate a defect in the nail matrix. Psoriasis can change the nail bed as the results in onycholysis, discoloration, splinter hemorrhage and subungual hyperkeratosis. The main treatment of psoriatic nails is using topical high- potent steroids however topical steroids are limited their ability to penetrate deep nail matrix or nail bed which are the main pathology. Use of such a treatment can lead to skin atrophy and report in the case of "Disappearing digits". Previous studies of steroid injection in the treatment of psoriatic nails show satisfactory results without any serious permanent adverse effects. At present, there is no comparison study between intralesional steroid and ultrapotent topical steroid for the treatment of psoriatic nails.

The purpose of the study is to evaluate the efficacy and safety of intralesional triamcinolone comparing to 0.05% clobetasol ointment in the treatment of psoriatic nails.

DETAILED DESCRIPTION:
Psoriasis is a chronic inflammatory disorder. The nails involvement has been reported up to 40% of psoriatic patients. Psoriatic nails can significantly affect a quality of life of patients. Psoriasis affects both nail matrix and nail bed. Pitting, leukonychia and red spots in lunula indicate a defect in the nail matrix. Psoriasis can change the nail bed as the results in onycholysis, discoloration, splinter hemorrhage and subungual hyperkeratosis. The main treatment of psoriatic nails is using topical high- potent steroids however topical steroids are limited their ability to penetrate deep nail matrix or nail bed which are the main pathology. Use of such a treatment can lead to skin atrophy and report in the case of "Disappearing digits". Previous studies of steroid injection in the treatment of psoriatic nails show satisfactory results without any serious permanent adverse effects. At present, there is no comparison study between intralesional steroid and ultrapotent topical steroid for the treatment of psoriatic nails.

The purpose of the study is to evaluate the efficacy and safety of intralesional triamcinolone comparing to 0.05% clobetasol ointment in the treatment of psoriatic nails.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged over 18 years old who have at least 3 psoriatic finger nails resembly severity

Exclusion Criteria:

1. Patients are receiving the systemic therapy of psoriasis
2. Patients discontinued the systemic therapy less than 3 months and topical therapy less than 1 month
3. Positive results for the microscopic study of fungus in finger nails
4. History of steroids or EMLA allergy
5. Pregnancy or nursing
6. Any skin infection at the site of the treatment
7. Human immunodeficiency virus subjects
8. History of malignancy or during the treatment of malignancy
9. Patients who have psychological disorder
10. Patients who have bleeding disorder or receiving anticoagulation drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-11; Primary Completion 2012-03 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Percent change in the NAPSI (Nail Psoriasis Severit Index) score of psoriatic nails after treatment with intralesional 0.1%triamcinolone injection vs.topical 0.05% clobetasol propionate ointment | 6 months
  1. To compare the percent change in the NAPSI (Nail Psoriasis Severity Index) score of Psoriatic nails after treatment with intralesional 0.1%triamcinolone injection vs.topical 0.05% clobetasol propionate ointment and controlled untreated group.

SECONDARY OUTCOMES:
adverse effects of the intralesional steroid injection and topical 0.05% clobetasol propionate ointment | 6 months
  Observe the possible adverse effects of the intralesional steroid injection and topical 0.05% clobetasol propionate ointment treatment for psoriatic nails.

CONTACTS AND LOCATIONS:
Overall Officials: Chanisada Wongpraparut, M.D., Principal Investigator — Siriraj Hospital
Locations (1):
- Siriraj Hospital, Bangkok, Bangkok, Thailand